CLINICAL TRIAL: NCT07095699
Title: An Exploratory, Parallel Controlled Study to Explore the Effectiveness of Intraoperative Margin Exploration Techniques for Adenocarcinoma of the Esophagogastric Junction
Brief Title: Intraoperative Margin Techniques for Esophagogastric Junction Adenocarcinoma: A Controlled Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Fenglin Liu, senior doctor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20250308
Record Dates: First submitted 2025-07-23; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-06

CONDITIONS: Adenocarcinoma of the Esophagogastric Junction
Keywords: AEG resection; fluorescent; microscope

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ES group (Experimental): ES-assisted surgery
  Interventions: Device: EndoSCell System
- FS Group (No Intervention): Frozen Section without ES scanning

INTERVENTIONS:
Device: EndoSCell System — EndoSCell Scaner (ES) is a new type of intraoperative cell-level fluorescence-guided imaging technology that can be used for direct and rapid intraoperative tissue cell interpretation. This technology uses a handheld cell microscope system to magnify local tissue by about 1280 times, and can perform rapid real-time scanning and imaging of in vivo or excised ex vivo tissue.
  Arms: ES group

SUMMARY:
The goal of this clinical trial is to learn if the EndoScell Scanner (ES) imaging system can accurately assess tumor-free surgical margins during surgery for adenocarcinoma of the esophagogastric junction (AEG), compared with standard frozen-section pathology.

The main questions it aims to answer are:

* Is ES non-inferior to intraoperative frozen-section pathology in identifying positive or negative tumor margins?
* Does ES shorten the time needed for margin assessment and reduce the number of additional tissue resections required?

Researchers will compare an ES-assisted surgical arm with a conventional frozen-section arm to see if ES improves margin accuracy, shortens operative time, and increases the rate of complete (R0) tumor removal.

Participants will

* undergo standard AEG resection with randomized assignment to either ES or frozen-section margin checks;
* allow collection of margin tissue samples for ES, frozen-section, and final paraffin pathology;
* attend routine follow-up visits for up to 2 years to monitor for local recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically diagnosed with adenocarcinoma of the esophagogastric junction (AEG):

Including patients with Siewert type II and III AEG; Including patients in cT1 stage (recommended esophageal resection margin distance ≥1.5cm) and cT2 and above (recommended esophageal resection margin distance ≥3cm);

* Plan to receive surgical resection of AEG;
* Patients voluntarily participated in this study and signed the informed consent form;

Exclusion Criteria:

* Patients who are allergic to methylene blue and fluorescein sodium;
* Patients with severe cardiovascular or circulatory system diseases and cannot tolerate surgery;
* Participated in other clinical trials of research drugs or devices in the past month;
* Unable to understand the test requirements or unable to complete the study follow-up plan;
* Pregnant and lactating women;
* Patients who are unable to complete follow-up due to mental illness, cognitive or emotional disorders;
* Subjects who are considered by the researchers to be unsuitable for participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy | intraoperative
  Using paraffin pathology as the gold standard, the accuracy of ES system and frozen pathology for AEG resection margin was evaluated: Accuracy Rate = true positive + true negative/total number of samples.

SECONDARY OUTCOMES:
Evaluation of R0 resection rate | 7days after the surgery
  The proportion of surgical resection specimens without residual tumor at the resection margin using paraffin pathology as the gold standard.
Positive margin rate | 7days after the surgery
  Using paraffin pathology as the gold standard, the proportion of ES interpretation as positive but frozen pathology showing negative
Evaluation of the actual resection margin distance during ES-assisted AEG | 7days after the surgery
  Evaluation of the actual resection margin distance during ES-assisted AEG
Evaluate the sensitivity, specificity, PPV, and NPV of ES technology | 7days after the surgery
  Evaluate the sensitivity, specificity, PPV, and NPV of ES technology
Evaluation of the consistency between ES technique and frozen pathology | 7days after the surgery
  Evaluation of the consistency between ES technique and frozen pathology
Postoperative recurrence: evaluate the anastomotic recurrence rate at 6, 12 months, and 2 years after surgery | 6, 12 months, and 2 years after surgery
  Postoperative recurrence: evaluate the anastomotic recurrence rate at 6, 12 months, and 2 years after surgery
Evaluation of the time efficiency of ES and frozen pathology | 7days after the surgery
  ES real-time interpretation time vs frozen pathology result time
Evaluate the number of timely adjustments to the resection range due to the interpretation of ES technology; | 7days after the surgery
  Evaluate the number of timely adjustments to the resection range due to the interpretation of ES technology;

OTHER OUTCOMES:
Accuracy of ES interpretation in different Siewert classifications (type II vs. type III) | 7days after the surgery
  Accuracy of ES interpretation in different Siewert classifications (type II vs. type III)

IPD SHARING:
Plan to Share IPD: Undecided